CLINICAL TRIAL: NCT06622889
Title: The Effectiveness of Interventions Targeting Self-Perception of Aging in Older Adults with Subjective Cognitive Decline
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng Li (Other)
Responsible Party: Sponsor-Investigator, Zheng Li, Professor, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUMCSON-2023-05
Record Dates: First submitted 2024-09-27; First posted 2024-10-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Subjective Cognitive Decline (SCD)
Keywords: Subjective Cognitive Decline; Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8-week intervention targeting self-perception of aging (Experimental): Participants in this condition will receive an 8-week intervention targeting self-perception of aging. Group sessions will be held at community health service centers, with one session per week, each lasting 45 to 60 minutes. Additionally, homework assignments will be supplemented, and researchers will provide additional remote support via WeChat.
  Interventions: Other: Multidomain Intervention Program
- Controls (No Intervention)

INTERVENTIONS:
Other: Multidomain Intervention Program — The intervention program aims to help older adults with subjective cognitive decline understand the aging process and adopt a positive attitude toward aging, highlighting age-related benefits. The sessions also provide emotion regulation techniques and stress-coping strategies to encourage proactive problem-solving and build confidence in handling challenges. By recalling positive life experiences, the program seeks to strengthen emotional connections, enhance the sense of belonging, and reconstruct a meaningful later life.
  Arms: 8-week intervention targeting self-perception of aging

SUMMARY:
Subjective cognitive decline (SCD) represents the initial clinical manifestation in the disease spectrum of Alzheimer's Disease (AD). It represents an essential stage for early prevention and treatment of cognitive impairment, making the SCD population an optimal target for prior intervention. This study aims to assess the feasibility and efficacy of an 8-week intervention targeting self-perception of aging in community-dwelling older adults with SCD.

DETAILED DESCRIPTION:
Dementia, especially Alzheimer's Disease (AD), is a major healthcare issue in aging populations. It not only threatens the physical and mental health of older adults but also imposes significant economic and caregiving burdens on families and society. As a preclinical stage of AD, subjective cognitive decline (SCD) is regarded as the optimal phase for early intervention in cognitive impairment. When confronted with the threats of physical, psychological, and social aging, older adults with SCD often hold negative perceptions and emotional responses toward their own aging. They tend to attribute physical decline and memory loss to normal aging processes, overlooking controllable factors, which poses potential risks to their future cognitive outcomes, such as accelerated cognitive decline, elevated dementia risk, and increased accumulation of AD biomarkers. This study is based on the Transactional Model of Stress and Coping (TMSC) and identifies the mechanisms through which self-perception of aging influences cognitive function in older adults with SCD. A comprehensive 8-week intervention program was developed to target these mechanisms. The 8-week intervention program aims to provide practical evidence for delaying cognitive decline in older adults with SCD by enhancing their positive perceptions of aging.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥60 years;
* residing in the community for 6 months at least;
* experiencing a consistent decline in self-reported cognitive abilities;
* having standard cognitive test performance in the normal range;
* willing to participate in this study.

Exclusion Criteria:

* having diagnosis of any neurological diseases including Parkinson's disease, brain tumor, cerebral infarction, encephalitis, epilepsy, etc.;
* having diagnosis of mental illness such as depression, anxiety, bipolar disorder, and schizophrenia;
* with history of substance abuse or addiction;
* with severe visual or hearing impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive Decline | Baseline (pre-intervention)，8 weeks (post-intervention)，and 16 weeks (follow-up)
  The 9-item Subjective Cognitive Decline Questionnaire (SCD-Q9) consists of 9 items. Higher scores indicate a greater likelihood of subjective cognitive impairment.

SECONDARY OUTCOMES:
Cognitive Function | Baseline (pre-intervention)，8 weeks (post-intervention)，and 16 weeks (follow-up)
  The Montreal Cognitive Assessment Beijing Version (MoCA-Beijing) encompasses multiple cognitive domains, including visuospatial execution ability, naming, memory and delayed recall, attention, language, abstraction, and orientation. The total score ranges from 0 to 30 points, and the higher the score, the better the overall cognitive function. Assessment tools of other cognitive domains will be used depending on the progress of the intervention program.
Self-perception of Aging | Baseline (pre-intervention)，8 weeks (post-intervention)，and 16 weeks (follow-up)
  The Chinese version of the Brief Aging Perceptions Questionnaire (B-APQ) comprises 17 items grouped into 5 dimensions. Participants rated their agreement on a Likert 5-point scale ranging from "strongly disagree" to "strongly agree" (1 to 5 scores). The total score ranges from 17 to 85 points, with higher scores indicating more negative self-perceived aging.
Perceived Stress | Baseline (pre-intervention)，8 weeks (post-intervention)，and 16 weeks (follow-up)
  The Chinese version of the Perceived Stress Scale (CPSS) will be used to measure individuals' perceived stress when facing stressful events. It consists of 14 items, with higher scores indicating higher level of perceived stress.
Coping Strategies | Baseline (pre-intervention)，8 weeks (post-intervention)，and 16 weeks (follow-up)
  The Simplified Coping Skill Questionnaire (SCSQ) includes two dimensions: positive coping and negative coping. Higher average scores in each dimension indicate a greater frequency of using that particular coping strategy.

OTHER OUTCOMES:
Satisfaction questionnaire | 8 weeks (post-intervention)
  The satisfaction questionnaire designed by the researchers will be used.
Compliance | 8 weeks (post-intervention)
  Percentage of participants who complete the whole intervention program, and the reasons for failure to comply
Acceptability interview | 8 weeks (post-intervention)
  After the end of the whole intervention, semi-structured interviews will be conducted with the subjects of the intervention group who volunteered to participate in the interview.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No